CLINICAL TRIAL: NCT06031922
Title: Comparing the Effectiveness and Cost-effectiveness of Conventional Mechanical Knees and Microprocessor-controlled Knees: a Prospective Cohort Study
Brief Title: Effectiveness and Cost-effectiveness of Lower Limb Prostheses
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Other Study IDs: 671860
Record Dates: First submitted 2023-08-23; First posted 2023-09-11 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Amputation; Prosthesis User; Prosthesis
Keywords: Effectiveness; transfemoral amputation; knee-disarticulation; Microprocessor controlled knee; prosthetic knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Microprocessor controlled knee — Microprocessor controlled knee

SUMMARY:
The goal of this observational study is to investigate the effectiveness of NMPKs versus MPKs in persons with an LLA in the standard healthcare system in the Netherlands taking all levels of the ICF model into account. Our main aim is to assess the effect of MPK use compared to NMPK use on walking distance, as this is one of the most used outcome variables in literature and thus enables comparison with previous studies. Our secondary aim is to investigate the effect of NMPKs versus MPKs on all ICF-levels: body structures and function, activities and participation.

Participants will be seen four times in a year. During these measurement moments they will:

* Perform two physical tests
* Fill out a set of questionnaires
* Wear an activity tracker for one week

DETAILED DESCRIPTION:
In this prospective cohort study the participants made use of two types of prosthetic knees; the CMK and MKP. A baseline measurement (T0) was performed while the participants were using their own CMK. One week later, they received the MPK to start a six week-trial. During this trial, they received 30 minutes of physical therapy twice a week. In the last week of the trial period, the measurements were performed again (T1). After the trial period, participants switched back to their CMK and after four weeks of getting used to that, the functional performance tests were repeated (T2). Nine months after the last measurement, and if the participant received a MPK, the measurements were repeated again (T3).

The measurements consisted of:

Physical tests:

* 6 minute walking test (6MWT)
* Timed up and Go test (TUGtest)

Questionnaires:

* Cost questionnaire
* Activities-Specific Balance Confidence Scale (ABC-NL)
* Utrecht Scale for Evaluation of Rehabilitation Participation (USER-P)
* Short Questionnaire to Assess Health-enhancing physical activity (SQUASH)
* Prosthesis Evaluation Questionnaire (PEQ)

Activity monitor:

* Activ8 professional. Worn for seven consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* At least one year post amputation
* Unilateral transfemoral amputation or knee-disarticulation
* Eligible for a trial on an MPK
* Able to read and write in Dutch
* Use a prosthesis with a socket

Exclusion Criteria:

* Bilateral amputation
* Osseointegration
* Previous experience with an MPK

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We included adult participants with a unilateral transfemoral amputation or knee-disarticulation who were using a prosthesis with a CMK, but were eligible for a trial on an MPK.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
6 Minute Walking Test (6MWT) | This test takes 6 minutes and is performed at T0 (week 1 after inclusion), T1 (week 7 after inclusion), T2 (week 12 after inclusion) and T3 (week 52 after inclusion)
  The 6-minute walk test is used to measure functional capacity. The maximum distance a participant can walk within 6 minutes is measured. The course can be 10, 30 or 50 meters. The participant can use their walking aid if needed.

SECONDARY OUTCOMES:
Short Questionnaire to Assess Health-enhancing physical activity (SQUASH) | Participants were asked to fill out the questionnaire at T0 (week 1 after inclusion), T1 (week 7 after inclusion) and T3 (week 52 after inclusion), with a normal/standard week for them in mind.
  The SQUASH is a questionnaire to measure physical activity [29]. The list is based on the Dutch Standard for Healthy Exercise [30]. This questionnaire contains 11 items to be completed by the participant. The SQUASH measures the frequency, duration and intensity of four different physical activities, namely: physical activity to and from work; household activities; activities at work; and physical activities performed in leisure time. The higher the score, the more time is spent on physical activities.
Timed Up and Go test (TUGtest) | This test is performed at T0 (week 1 after inclusion), T1 (week 7 after inclusion), T2 (week 12 after inclusion) and T3 (week 52 after inclusion). It can take up to three minutes.
  The Timed Up & Go test (TUG) measures the time it takes the participant to get up from a chair, walk 3 meters comfortably, turn around, walk back and sit down. Participants are allowed to use their walking aids, but no physical assistance or encouragement should be given.
Activities-Specific Balance Confidence Scale Nederlands (ABC-NL) | Participants were asked to fill out the questionnaire at T0 (week 1 after inclusion), T1 (week 7 after inclusion) and T3 (week 52 after inclusion), based on their current situation that day.
  The Activities-Specific Balance Confidence (ABC) Scale is a questionnaire consisting of 16 items. For each item/activity, the patient should indicate how much confidence he/she has in not falling or losing balance when performing them. Each question is scored from 0% to 100% confidence. The activities described take place both indoors and outdoors and are diverse. A high score corresponds to a lot of confidence to perform the activity.
Cost-questionnaire | At T0 (week 1 after inclusion) and T3 (week 52 after inclusion), participants were asked to fill out the questionnaire over a retrospective period of six months.
  To get insight in the costs, two existing questionnaires were combined: the Productivity Cost Questionnaire (iPCQ) and the Medical Consumption Questionnaire (iMCQ).
  The iMCQ is used to measure medical consumption. It includes questions related to the number of appointments with health care providers. The iPCQ measures and values productivity losses. It looks at absenteeism, presenteeism, productivity losses and unpaid work. As this study focussed on costs related to lower limb prostheses, questions about appointments with a dietician and speech therapist, and trips to the emergency room were replaced with questions about the type of prosthesis and the number of appointments with their prosthetist. Finally, questions about personal costs related to the acquisition and repairs of the prosthesis, as well as personal expenses were added.
Prosthesis Evaluation Questionnaire (PEQ) | Participants were asked to fill out the questionnaire at T0 (week 1 after inclusion), T1 (week 7 after inclusion) and T3 (week 52 after inclusion) over a retrospective period of four weeks.
  The PEQ is a reliable and valid self-report questionnaire to evaluate prosthesis and prosthesis-related quality of life. Questions are divided into nine subscales (ambulation, perceived response, sounds, appearance, residual limb health, utility, frustration, social burden and well-being) and several separate questions related to pain, satisfaction, transfers, prosthetic care, self-efficacy and importance. Most questions are scored on a visual analogue scale (VAS) from 0-100. Some questions about the frequency of certain problems (e.g. pain in residual limb or back) are multiple choice. A higher score on this questionnaire is linked to a more positive outcome.
Utrecht Scale for Evaluation of Rehabilitation Participation (USER-P) | Participants were asked to fill out the questionnaire at T0 (week 1 after inclusion), T1 (week 7 after inclusion) and T3 (week 52 after inclusion) over a retrospective period of four weeks.
  This questionnaire is used to rate objective and subjective participation. It is composed of 31 items, divided over three scales: 1) frequency: 1a. how much time the participant spends on work, study and household per week, rated on a scale from 0 (not at all) up to 5 (36 hours or more) and 1b. how often the participant partakes in certain activities per week, scored from 0 (not at all) up to 5 (19 times or more); 2) restrictions: whether the participant experiences limitations in daily life and whether they could do certain activities with or without help, scored from 0 (not possible at all) to 3 (independent without difficulty); and 3) satisfaction: how satisfied the participant is with different aspects of daily life, scored on a range from 0 (very dissatisfied) to 4 (very satisfied).
Activity tracking for physical activity (Activ8) | The activity tracker was worn 24 hours a day for 7 days straight.
  The Active 8 professional activity monitor was used to register walking during one full week. The activity monitor was placed by the physical therapist on the thigh of the non-affected side of the participant. During the week, the participant was asked to fill out a short diary with the time they got up and went to bed; whether they had worn the monitor for the full 24 hours; whether they had done any physical activity that wasn't in their usual day-to-day routine; and if so during what time that activity was performed.

CONTACTS AND LOCATIONS:
Locations (9):
- Netherlands (9):
  - Revant medisch specialistische revalidatie, Breda
  - Revalidatiecentrum Roessingh, Enschede
  - Revant medisch specialistische revalidatie | Lindenhof, Goes
  - University Medical Center Groningen, Groningen
  - Adelante zorggroep, Hoensbroek
  - Rijndam Revalidatie, Rotterdam
  - De Hoogstraat Revalidatie, Utrecht
  - Heliomare Centrum voor Specialistische Revalidatie, Wijk aan Zee
  - Vogellanden, centrum voor medisch specialistische revalidatie, bijzondere tandheelkunde en gezonde leefstijl, Zwolle

IPD SHARING:
Plan to Share IPD: Undecided